CLINICAL TRIAL: NCT06407622
Title: The Effect of Foot Reflexology on Pain Intensity, Sleep Quality and Bowel Functions in Patients Undergoing Appendectomy Surgery
Brief Title: The Effect of Foot Reflexology on Patients Undergoing Appendectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Buket Köse Çetinalp, Nurse, Bartın Unıversity
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: BartınU-SBF-BKÇ-01
Record Dates: First submitted 2024-02-02; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Nursing; Pain; Reflexology; Abdominal Pain; Sleep Quality; Bowel Functions; Appendectomy
Keywords: Nursing; Pain; Reflexology; Abdominal Pain; Sleep Quality; Bowel Functions; Appendectomy
MeSH Terms: conditions — Pain; Abdominal Pain; Sleep Initiation and Maintenance Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: The thesis study was planned as a randomized controlled experimental study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients undergoing appendectomy surgery who received foot reflexology (Experimental): The study will be carried out with 120 patients hospitalized after appendectomy surgery in the surgical clinic of Bartın State Hospital. In the postoperative period, patients will be divided into experimental (n = 60) and control (n = 60) groups by block randomization with a computer-aided program.
  Interventions: Other: Foot Reflexology
- Patients who underwent appendectomy surgery without foot reflexology (No Intervention): The study will be carried out with 120 patients hospitalized after appendectomy surgery in the surgical clinic of Bartın State Hospital. In the postoperative period, patients will be divided into experimental (n = 60) and control (n = 60) groups by block randomization with a computer-aided program.

INTERVENTIONS:
Other: Foot Reflexology — In previous studies, no study was found investigating the effect of foot reflexology on sleep quality and bowel functions in patients undergoing surgical intervention. This study is thought to be the first to evaluate the effect of foot reflexology on sleep quality and bowel functions in surgical patients. In this respect, it is a study that will contribute to the literature.
  Other Names: Foot; Reflexology
  Arms: Patients undergoing appendectomy surgery who received foot reflexology

SUMMARY:
Pain is an unpleasant experience that can negatively affect all aspects of the patients life and lead to a decrease in quality of life. Pain can also be encountered as a reason for a surgical intervention. For this reason, it has become one of the most common problems experienced by patients in the postoperative period. Pain management is a universal requirement in health care and is of great importance for patients. If the pain is not managed well in the postoperative period, it may cause some complications in the patient. If pain is controlled, early discharge of the patient, lower healthcare costs and increased patient satisfaction are achieved. In terms of providing effective pain control, it is provided by nurses, who are health professionals, to spend more time with the patient, to lead the patient in pain management and to analyze the results. The aim of the thesis study is to evaluate the effect of foot reflexology on pain intensity, sleep quality and bowel functions in patients who have undergone appendectomy surgery.

DETAILED DESCRIPTION:
Optimal management of postoperative pain is associated with reduced morbidity and faster recovery times, as well as improved physical function and quality of life. Despite efforts to minimize postoperative pain, 61% of outpatients still experience moderate/extreme pain upon discharge. Pain management is an important aspect of patient care, and nurses play an important role in providing pain assessment and treatment in the acute care setting. The use of non-pharmacological pain relief techniques has been found to be effective with fewer side effects and complications. Reflexology, one of the types of complementary and alternative medicine, has begun to be used as a nursing intervention along with modern medicine as a non-pharmacological method. When the investigators look at the past years; The effects of foot reflexology on pain intensity, nausea, anxiety, delirium, and hemodynamic parameters were investigated. The studies conducted include cancer patients, burn patients, intensive care patients and dialysis patients. However, in previous studies, no study was found investigating the effect of foot reflexology on sleep quality and bowel functions in patients undergoing surgical intervention. This study is thought to be the first to evaluate the effect of foot reflexology on sleep quality and bowel functions in surgical patients. In this respect, it is a study that will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* • 18 years and over,

  * Having undergone appendectomy surgery,
  * No complications such as bleeding, nausea or vomiting after appendectomy surgery,
  * Not using patient-controlled analgesia for postoperative pain control,
  * Pain score ≥4 according to the Visual Analog Scale,
  * No hypertension problems,
  * Able to speak and understand Turkish
  * No visual or auditory problems,
  * No diagnosed psychiatric problems,
  * No diagnosed bowel problems,
  * Do not have infectious skin diseases on their feet (such as zoster, fungus, warts, eczema),
  * Patients who do not have deep vein thrombosis, tombophlebitis, any fracture, neuropathy, osteomyelitis, osteoporosis, or ligament injury in their feet or legs,
  * Volunteer patients will be included.

Exclusion Criteria:

* • Complications developed after appendectomy surgery,

  * Pain score <4 according to the Visual Analog Scale,
  * Those with hypertension problems,
  * Unable to communicate,
  * Having visual or auditory problems,
  * Having a diagnosed psychiatric problem,
  * Having a diagnosed bowel problem,
  * Those with infectious skin diseases on their feet (such as zoster, fungus, warts, eczema),
  * Patients with deep vein thrombosis, tombophlebitis, any fracture, neuropathy, osteomyelitis, osteoporosis, ligament injury in the foot and leg,
  * Non-voluntary patients will be excluded from the scope.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
The Effect of Foot Reflexology on Pain Intensity | initial postoperative evaluation, 1st hour and 3rd hour
  In this study, foot reflexology will be applied to patients who have undergone appendectomy surgery. After this reflexology, patients' pain intensity will be evaluated. When the patients come out of appendectomy surgery, their pain will be evaluated with visual analog scale(VAS). Then, no intervention will be applied to the control group. Foot reflexology massage will be applied to the patients in the intervention group at the 1st hour postoperatively and pain values will be measured with VAS at 5 minutes, 30 minutes and 60 minutes after this application. At the 3rd hour postoperatively, reflexology massage will be performed for the 2nd time and pain intensity will be evaluated with VAS at 5 minutes, 30 minutes and 60 minutes after the re-massage.
  VAS pain score is evaluated as "no pain" (score=0) and "worst pain" (score=10). score <3 is reported as mild pain, 3-6 as mild-moderate pain and >6 as moderate-severe pain.
The Effect of Foot Reflexology on Sleep Quality | 24 hours after surgery
  After appendectomy surgery, no intervention will be applied to the control group, while foot reflexology will be applied to the intervention group at the 1st and 3rd hour after surgery. At 24 hours, the sleep quality of the intervention and control group patients will be evaluated with the Richard Cambple Sleep Scale.
  Richard Campbell sleep scale consists of 6 items. Total scoring is based on the first 5 items. Each item is evaluated on a scale of 0-100 with the visual analog scale technique. A score of 0-25 on the scale indicates very poor sleep and 76-100 indicates very good sleep.
The Effect of Foot Reflexology on Bowel Function | initial postoperative evaluation, 1st hour and 3rd hour
  After appendectomy, bowel functions of the control and intervention groups will be evaluated. Afterwards, foot reflexology will be applied to the intervention group at the 1st and 3rd hour and their bowel functions will be evaluated on the bowel monitoring form. The control group will be evaluated at the 1st hour and 3rd hour after surgery without any intervention. Bowel functions will be recorded on the bowel function monitoring form created by the researcher. This form includes parameters such as the time of the first flatulence, the time of the first defecation, the time of oral feeding, and the time of the first mobilization.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim ÇELİK, Prof, Study Director — Bartın University Health Science Faculty
Locations (1):
- Bartın University, Bartın, Centrical, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zeidabadinejad S, Mangolian Shahrbabaki P, Dehghan M. Effect of Foot Reflexology on Sexual Function of Patients under Hemodialysis: A Randomized Parallel Controlled Clinical Trial. Evid Based Complement Alternat Med. 2021 Oct 21;2021:8553549. doi: 10.1155/2021/8553549. eCollection 2021. PMID 34721645
- [Result] Wang WL, Hung HY, Chen YR, Chen KH, Yang SN, Chu CM, Chan YY. Effect of Foot Reflexology Intervention on Depression, Anxiety, and Sleep Quality in Adults: A Meta-Analysis and Metaregression of Randomized Controlled Trials. Evid Based Complement Alternat Med. 2020 Sep 15;2020:2654353. doi: 10.1155/2020/2654353. eCollection 2020. PMID 33014101
- [Result] Taheri H, Naseri-Salahshour V, Abedi A, Sajadi M. Comparing the Effect of Foot and Hand Reflexology on Pain Severity after Appendectomy: A Randomized Clinical Trial. Iran J Nurs Midwifery Res. 2019 Nov 7;24(6):451-456. doi: 10.4103/ijnmr.IJNMR_85_18. eCollection 2019 Nov-Dec. PMID 31772920
- [Result] Samuel SR, Gururaj R, Kumar KV, Vira P, Saxena PUP, Keogh JWL. Randomized control trial evidence for the benefits of massage and relaxation therapy on sleep in cancer survivors-a systematic review. J Cancer Surviv. 2021 Oct;15(5):799-810. doi: 10.1007/s11764-020-00972-x. Epub 2020 Dec 2. PMID 33269414
- [Result] Samarehfekri A, Dehghan M, Arab M, Ebadzadeh MR. Effect of Foot Reflexology on Pain, Fatigue, and Quality of Sleep after Kidney Transplantation Surgery: A Parallel Randomized Controlled Trial. Evid Based Complement Alternat Med. 2020 Aug 1;2020:5095071. doi: 10.1155/2020/5095071. eCollection 2020. PMID 32831868
- [Result] Rejeh N, Tadrisi SD, Yazdani S, Saatchi K, Vaismoradi M. The Effect of Hand Reflexology Massage on Pain and Fatigue in Patients after Coronary Angiography: A Randomized Controlled Clinical Trial. Nurs Res Pract. 2020 Aug 29;2020:8386167. doi: 10.1155/2020/8386167. eCollection 2020. PMID 32908698
- [Result] Paul RW, Szukics PF, Brutico J, Tjoumakaris FP, Freedman KB. Postoperative Multimodal Pain Management and Opioid Consumption in Arthroscopy Clinical Trials: A Systematic Review. Arthrosc Sports Med Rehabil. 2021 Dec 17;4(2):e721-e746. doi: 10.1016/j.asmr.2021.09.011. eCollection 2022 Apr. PMID 35494281
- [Result] Mwanza E, Gwisai RD, Munemo C. Knowledge on Nonpharmacological Methods of Pain Management among Nurses at Bindura Hospital, Zimbabwe. Pain Res Treat. 2019 Jan 1;2019:2703579. doi: 10.1155/2019/2703579. eCollection 2019. PMID 30693106
- [Result] Koffel E, Kats AM, Kroenke K, Bair MJ, Gravely A, DeRonne B, Donaldson MT, Goldsmith ES, Noorbaloochi S, Krebs EE. Sleep Disturbance Predicts Less Improvement in Pain Outcomes: Secondary Analysis of the SPACE Randomized Clinical Trial. Pain Med. 2020 Jun 1;21(6):1162-1167. doi: 10.1093/pm/pnz221. PMID 31529104
- [Result] Gordon-Williams R, Trigo A, Bassett P, Williams A, Cone S, Lees M, Brandner B. An Interactive Pain Application (MServ) Improves Postoperative Pain Management. Pain Res Manag. 2021 Apr 2;2021:8898170. doi: 10.1155/2021/8898170. eCollection 2021. PMID 33868524
- [Result] Ghanbari A, Shahrbabaki PM, Dehghan M, Mardanparvar H, Abadi EKD, Emami A, Sarikhani-Khorrami E. Comparison of the Effect of Reflexology and Swedish Massage on Restless Legs Syndrome and Sleep Quality in Patients Undergoing Hemodialysis: a Randomized Clinical Trial. Int J Ther Massage Bodywork. 2022 Jun 1;15(2):1-13. doi: 10.3822/ijtmb.v15i2.705. eCollection 2022 Jun. PMID 35686176
- [Result] Fazlollah A, Babatabar Darzi H, Heidaranlu E, Moradian ST. The effect of foot reflexology massage on delirium and sleep quality following cardiac surgery: A randomized clinical trial. Complement Ther Med. 2021 Aug;60:102738. doi: 10.1016/j.ctim.2021.102738. Epub 2021 May 21. PMID 34029674
- [Result] Blackburn L, Hill C, Lindsey AL, Sinnott LT, Thompson K, Quick A. Effect of Foot Reflexology and Aromatherapy on Anxiety and Pain During Brachytherapy for Cervical Cancer. Oncol Nurs Forum. 2021 May 1;48(3):265-276. doi: 10.1188/21.ONF.265-276. PMID 33855996
- [Result] Alinia-Najjar R, Bagheri-Nesami M, Shorofi SA, Mousavinasab SN, Saatchi K. The effect of foot reflexology massage on burn-specific pain anxiety and sleep quality and quantity of patients hospitalized in the burn intensive care unit (ICU). Burns. 2020 Dec;46(8):1942-1951. doi: 10.1016/j.burns.2020.04.035. Epub 2020 May 19. PMID 32873443